CLINICAL TRIAL: NCT05198973
Title: Bumblebee Breath Effect on Tinnitus in Older Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: P.T.REC/012/003456
Record Dates: First submitted 2021-12-05; First posted 2022-01-20 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Tinnitus, Subjective
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bumblebee Breath group (Experimental): Bumblebee Breath starts by finding a relaxed, supported posture, either laying supine or in seated and then bringing the minds attention to the space between the eyebrows (or third eye in yoga terms). With the eyes close the thumbs are placed over the tragus of the ears, the first finger gently rests on eye lids, middle finger touches the sides of the nose and then the index and pinkie rest just above and below the closed lips. Next, a sound is created by inhaling deeply through the nose and exhaling with a low-pitched humming sound. The result sounds very much like a bee buzzing to the person performing the breath and a sensation of vibration is experienced inside the head and over the face. this group will be 28 patients to receive half an hour daily for ( 1 month)
  Interventions: Behavioral: Bumblebee Breath
- control group (No Intervention): this group (28 patients) will receive no training

INTERVENTIONS:
Behavioral: Bumblebee Breath — Bumblebee Breath starts by finding a relaxed, supported posture, either laying supine or in seated and then bringing the minds attention to the space between the eyebrows (or third eye in yoga terms). With the eyes close the thumbs are placed over the tragus of the ears, the first finger gently rests on eye lids, middle finger touches the sides of the nose and then the index and pinkie rest just above and below the closed lips. Next, a sound is created by inhaling deeply through the nose and exhaling with a low-pitched humming sound. The result sounds very much like a bee buzzing to the person performing the breath and a sensation of vibration is experienced inside the head and over the face.
  this will applied half an hour daily for ( 1 month)
  Arms: Bumblebee Breath group

SUMMARY:
Tinnitus is a condition in which the person hears sound, which isn't coming from the external environment, often, described as ringing in the ears.

Patients describe the condition as an annoyance and disturbance and in turn this correlates with increased levels of anxiety and depression. Currently, there is no single effective treatment for tinnitus so research continues to look for new ways to treat and manage the condition.

Bumblebee Breath starts by finding a relaxed, supported posture, either laying supine or in seated and then bringing the minds attention to the space between the eyebrows (or third eye in yoga terms). With the eyes close the thumbs are placed over the tragus of the ears, the first finger gently rests on eye lids, middle finger touches the sides of the nose and then the index and pinkie rest just above and below the closed lips. Next, a sound is created by inhaling deeply through the nose and exhaling with a low-pitched humming sound. The result sounds very much like a bee buzzing to the person performing the breath and a sensation of vibration is experienced inside the head and over the face. this study is designed to assess Bumblebee Breath on tinnitus.

DETAILED DESCRIPTION:
two groups (28 for each) will included. One tinnitus group will receive half an hour of Bumblebee Breath training (daily) for one month. The second one will receive nothing

ELIGIBILITY:
Inclusion Criteria:

* elderly males and females
* Tinnitus complaints

Exclusion Criteria:

* cardio(respiratory) symptoms, any local (within ear) problem(s).

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — self-representation of gender identity.
Enrollment: 56 (Estimated)
Dates: Start 2021-11-08 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Tinnitus Handicap Inventory | week 4
  life-quality inquiry in tinnitus subjects (if its score decreases, it means tinnitus improvement)

SECONDARY OUTCOMES:
visual analogue scale for tinnitus annoyance | week 4
  measures of tinnitus annoyance
visual analogue scale for tinnitus loudness | week 4
  measures of tinnitus loudness
pulse rate | week 4
  autonomic-status assessment
respiratory rate | week 4
  autonomic-status assessment
systolic blood pressure | week 4
  force of blood during ventricular contraction
diastolic blood pressure | week 4
  force of blood during ventricular relaxation

CONTACTS AND LOCATIONS:
Overall Officials: Ali Ismail, lecturer, Principal Investigator — Cairo University
Locations (1):
- Cairo Unoversity, Giza, Egypt